CLINICAL TRIAL: NCT00131729
Title: Electronic Recording of Compliance With Occlusion Therapy for Amblyopia: 1 Effects of Patient Education on Compliance 2 Predictors for Non-Compliance
Brief Title: Electronic Recording of Compliance With Occlusion Therapy for Amblyopia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Albert von Metzler Foundation (Other); Augenstern Association, Germany (Unknown); Edith von Heyden Foundation, Germany (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2300.0020
Record Dates: First submitted 2005-08-18; First posted 2005-08-19 (Estimated); Last update posted 2006-03-20 (Estimated); Status verified 2006-03

CONDITIONS: Amblyopia
Keywords: Amblyopia; Occlusion therapy; Compliance; Risk factors
MeSH Terms: conditions — Amblyopia; Patient Compliance

INTERVENTIONS:
Behavioral: Educational programme

SUMMARY:
The purpose of this study was to determine whether compliance with occlusion therapy for amblyopia could be improved and, secondly, if risk factors for non-compliance could be identified.

DETAILED DESCRIPTION:
Non-compliance is a limiting factor for success of occlusion therapy for amblyopia (lazy eye) in childhood. It is responsible for approximately 1% of the adult population being unable to read with the amblyopic eye. The researchers used electronic monitoring of compliance to investigate predictors and a remedy for non-compliance.

Methods: In a prospective randomised controlled trial, compliance was measured for one week every three months during 30 months in newly diagnosed amblyopic children in The Hague, Frankfurt and Leicester. The family's social-economic and ethnic background was assessed through a questionnaire. Children were randomised to receive either an educational cartoon story explaining, without text, the rationale for treatment to the child with reward stickers and an information sheet, or a picture to colour. All received standard orthoptic care by a treating orthoptist, who was unaware of the randomisation. The electronic device and educational programme were distributed via home-visits by researchers. The primary outcome measure was percentage of compliance (realised/prescribed occlusion time). The secondary outcome measure was influence of social-economic, ethnic and clinical factors on compliance.

ELIGIBILITY:
Inclusion Criteria:

* All newly diagnosed amblyopic children with an inter-ocular difference in visual acuity of at least 0.2 logMAR, strabismus and/or anisometropia or deprivation (e.g. cataract)

Exclusion Criteria:

* Previous treatment for amblyopia
* Neurological disorder
* Medication
* Other eye disorder
* Decreased visual acuity caused by brain damage or trauma

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2001-07; Study Completion 2005-12

PRIMARY OUTCOMES:
Percentage of compliance (realised/prescribed occlusion time) in the intervention and control group

SECONDARY OUTCOMES:
Secondary outcome measure was influence of social-economic, ethnic and clinical factors on compliance

CONTACTS AND LOCATIONS:
Overall Officials: Huibert J Simonsz, MD, PhD, Study Chair — ErasmusMC, Department of Ophthalmology
Locations (2):
- Universitäts-Augenklinik Frankfurt, Frankfurt am Main, Germany
- Leicester Royal Infirmary; Dept. of Ophthalmology, Leicester, United Kingdom